CLINICAL TRIAL: NCT02027597
Title: Improving Oral Health With Serious Games
Acronym: AOTSM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Jacqueline E. Pickrell, Acting Assistant Professor, Oral Health Sciences, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 35095-EB; 5R44DE019043-02 (NIH)
Record Dates: First submitted 2014-01-02; First posted 2014-01-06 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2014-01

CONDITIONS: Caries; Tooth Decay; Cavities; Gingivitis
Keywords: video games; oral health; social cognitive theory; behavior change; randomized trial; growth modeling; minority; gender
MeSH Terms: conditions — Dental Caries; Gingivitis; Coitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Video Game Treatment (Experimental): This group received the AOTSM game experience followed by additional oral health information. They did not receive any follow-up treatment after the exhibit.
  Interventions: Other: Attack of the S. Mutans
- Control (Active Comparator): Instead of playing Attack of the S. Mutans!, children in the control group attended a 90 minute classroom session about virtual reality applications for relieving pain and for therapy. This content was unrelated to oral health.
  Interventions: Other: SnowWorld
- Video Game Treatment Plus Follow-Up (Experimental): Children assigned to the Treatment-Plus conditions not only had the Attack of the S. Mutans video game experience, but also gained access to an educational website that reinforced the exhibit's teachings two months later. These students received a special login and password in the mail and were instructed to visit the site before completing their next questionnaire.
  Interventions: Other: Attack of the S. Mutans; Other: Follow-up

INTERVENTIONS:
Other: Attack of the S. Mutans — A research assistant led groups of students through the Attack of the S. Mutans exhibit. All participants played all the games and viewed all the graphical content of the exhibit.
  Other Names: AOTSM
  Arms: Video Game Treatment; Video Game Treatment Plus Follow-Up
Other: Follow-up — This group experienced the Attack of the S. Mutans! exhibit and 3 doses of follow-up booster content at a web site.
  Arms: Video Game Treatment Plus Follow-Up
Other: SnowWorld — SnowWorld is a 3D first-person-shooter game developed by Firsthand Technology. In SnowWorld, the player shoots snowballs at penguins, polar bears, and other features of a frozen landscape. The game is designed to help burn victims cope with pain, and has no oral health messages.
  Arms: Control

SUMMARY:
This study investigated if computer games can be effective at changing the way children take care of their teeth. We a museum exhibit with 3D virtual reality games called "Attack of the S. Mutans!" Our hypothesis was that children who played the games and visited the exhibit would show improved attitudes about oral health, which would translate into improved brushing and self-care habits.

In this randomized controlled study with school children aged 8-12, we compared the outcomes for three groups: Group 1) Visited Attack of the S. Mutans!; Group 2) Experienced a hands-on classroom presentation about virtual reality being used for healthcare; Group 3) Received no-treatment.

ELIGIBILITY:
Inclusion Criteria:

For participation in the study, enrollment criteria are as follows: 1) a dentist's diagnosis of tooth decay, or restorative dental work in the previous year; and 2) Parents or guardians provide usable baseline data, including contact information for follow-up questionnaires.

Exclusion Criteria:

None

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 161 (Actual)
Dates: Start 2008-10; Primary Completion 2010-12 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Self-Efficacy | 8 months post treatment
  Follow-up surveys were conducted at 3 points after the intervention for all groups. The survey included questions about the children's attitudes (self-efficacy) toward oral health and taking care of their teeth. Surveys were paper-pencil self-reports from both parents and children. Items were drawn from Morowatisharifabad and Shirazi, (2007) and adapted for ease of understanding for English speaking children.

SECONDARY OUTCOMES:
Self-care behavior | 8 months post treatment
  Separate surveys of children and their parents were conducted at 3 points after the intervention all groups. The survey included questions about how often and how well the children took care of their teeth.

OTHER OUTCOMES:
Oral health literacy | 8 months post treatment
  we assessed children's oral health knowledge in two ways. First, children reported their overall oral health knowledge using three-point rating scales (=not really to 3=mostly) to respond to six items, including, "By brushing and flossing my teeth, I am less susceptible to tooth decay." Negatively worded items were reverse-coded, and the estimated internal consistency (Cronbach's alpha) of the pre-game survey was.49. Second, children indicated their brushing knowledge using five-point rating scales (1=strongly disagree to 5=strongly agree) to respond to four items, including "Tooth brushing gets rid of bad breath."

CONTACTS AND LOCATIONS:
Overall Officials: Howard A Rose, M.Ed., Principal Investigator — Firsthand Technology; Ari J Hollander, MSE, Principal Investigator — Firsthand Technology
Locations (1):
- Firsthand Technology Inc., Seattle, Washington, United States

REFERENCES:
- See also: Web site for Firsthand Technology, creators of Attack of the S. Mutans! — http://www.firsthand.com